CLINICAL TRIAL: NCT03611959
Title: Transformed Waldenström Macroglobulinaemia: Clinical Presentation and Outcome. A Multi-institutional Retrospective Study of 77 Cases From the French Innovative Leukemia Organization (FILO)
Brief Title: Transformed Waldenström Macroglobulineamia
Acronym: tWM
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2017Ao004
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Transformed Waldenström Macroglobulineamia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non Applicable

SUMMARY:
Histological transformation to diffuse large B-cell lymphoma is a rare complication which may occur in Waldenstrom macroglobulinemia. In this multicenter study, we retrospectively analyzed the clinico-biological features, therapy, outcomes and prognostic factors in 77 Waldenstrom macroglobulinemia patients with biopsy-proven transformation to diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Histological transformation to diffuse large B-cell lymphoma is a rare complication which may occur in Waldenstrom macroglobulinemia. In this multicenter study, we retrospectively analyzed the clinico-biological features, therapy, outcomes and prognostic factors in 77 Waldenstrom macroglobulinemia (WM) patients with biopsy-proven transformation to diffuse large B-cell lymphoma (DLBCL).

We retrospectively searched the databases of French and Belgian centers for patients older than 18 years diagnosed with WM and a concurrent or sequential diagnosis of DLBCL between 1995 and 2016. Nineteen centers belonging to the French Innovative Leukemia Organization (FILO) group participated in this study. Patients with a diagnosis of indolent lymphoma other than WM were excluded. The diagnosis of WM was based on criteria established in the Second International Workshop on WM. Clinical, biological data and prognostic scores were recorded. Quantitative variables were expressed as median and range and qualitative variables as number and percentages. Multivariate analyses using cox proportional hazard model were conducted to investigate the factors independently related to progression-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years diagnosed with Waldenstrom macroglobulineamia and a concurrent or sequential diagnosis of diffuse large B-cell lymphoma between 1995 and 2016

Exclusion Criteria:

* Patients with a diagnosis of indolent lymphoma other than Waldenstrom macroglobulineamia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years diagnosed with Waldenstrom macroglobulineamia and a concurrent or sequential diagnosis of diffuse large B-cell lymphoma between 1995 and 2016 were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 1995-01 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Description of clinical and biological features, therapeutic approaches, and clinical outcomes of patients with transformed Waldenstrom macroglobulineamia | 21 years

SECONDARY OUTCOMES:
Prognostic factor of progression-free survival (the time from diagnosis of histological transformation until progression, death from any cause or last follow-up) | 21 years
Prognostic factor of overall survival (the time from diagnosis of histological transformation until death from any cause or last follow-up) | 21 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Durot E, Tomowiak C, Michallet AS, Dupuis J, Hivert B, Lepretre S, Toussaint E, Godet S, Merabet F, Van Den Neste E, Ivanoff S, Roussel X, Zini JM, Regny C, Lemal R, Sutton L, Perrot A, Le Du K, Kanagaratnam L, Morel P, Leblond V, Delmer A. Transformed Waldenstrom macroglobulinaemia: clinical presentation and outcome. A multi-institutional retrospective study of 77 cases from the French Innovative Leukemia Organization (FILO). Br J Haematol. 2017 Nov;179(3):439-448. doi: 10.1111/bjh.14881. Epub 2017 Aug 2. PMID 28770576